CLINICAL TRIAL: NCT00951028
Title: Efficacy of CBT for Adherence and Depression in HIV Care Settings
Brief Title: Therapy Targeting Depression and HIV Treatment Adherence (The TRIAD Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven A. Safren, Director, Behavioral Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH084757 (NIH); R01MH084757 (NIH); 1R01MH084757-01A1 (NIH); DAHBR 9A-ASGA
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: HIV; Depression; HIV Infections
Keywords: Adherence
MeSH Terms: conditions — Depression; HIV Infections | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Enhanced treatment as usual (Active Comparator): Participants will receive the life-steps intervention and treatment as usual.
  Interventions: Behavioral: Life-steps adherence treatment
- CBT for adherence and depression (CBT-AD) (Experimental): Participants will receive the life-steps and CBT-AD interventions.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT) for adherence and depression (CBT-AD); Behavioral: Life-steps adherence treatment
- ISP for adherence and depression (ISP-AD) (Active Comparator): Participants will receive the life-steps and ISP-AD interventions.
  Interventions: Behavioral: Life-steps adherence treatment; Behavioral: Information and supportive psychotherapy (ISP) for adherence and depression (ISP-AD)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) for adherence and depression (CBT-AD) — 12 therapy sessions delivered over 4 months, using cognitive behavioral strategies to target depressive symptoms and adherence to HIV medications
  Arms: CBT for adherence and depression (CBT-AD)
Behavioral: Life-steps adherence treatment — Single-session adherence treatment that targets informational, problem solving, and cognitive-behavioral steps geared toward improving HIV medication adherence and self-management
Behavioral: Information and supportive psychotherapy (ISP) for adherence and depression (ISP-AD) — 12 therapy sessions delivered over 4 months, providing education and support that target depressive symptoms and adherence to HIV medications.
  Arms: ISP for adherence and depression (ISP-AD)

SUMMARY:
This study will test a therapy for both helping people adhere to their HIV medication regimens and treating them for depression.

DETAILED DESCRIPTION:
People infected with HIV are more likely to suffer from depression than those not infected, with studies finding anywhere from 20% to 50% of HIV-infected individuals having significant depressive symptoms. Depression, in addition to causing persistent sadness and inability to feel pleasure, is related to a lack of HIV treatment adherence. Treatment adherence (making sure to take every pill as prescribed by doctors) is critically important to successful treatment of HIV, because missing even a few doses gives the HIV virus an opportunity to develop immunity to the medication. Poor adherence is related to worse medical outcomes, but even a small, 10% improvement rate in adherence may improve these outcomes. This study will test the efficacy of cognitive behavioral therapy (CBT) that addresses both depression and treatment adherence for HIV-infected people.

Participation in this study will last 1 year, including follow-up visits. All participants will complete an initial one-visit intervention addressing treatment adherence. Then after 2 weeks, participants will be randomly assigned to one of three conditions: CBT for HIV medication adherence and depression (CBT-AD), information and supportive psychotherapy for HIV medication adherence and depression (ISP-AD), or enhanced treatment as usual (ETAU). Participants receiving CBT-AD and ISP-AD will complete 12 therapy sessions over 4 months and will be asked to report any changes to their psychological or HIV treatments. CBT-AD will involve learning to identify and change problematic patterns of thought and behavior, while ISP-AD will involve education and supportive psychotherapy. Participants receiving ETAU will receive only the initial session on HIV medication adherence and will be asked about their psychological and HIV treatment every other week for 4 months.

Major study assessments will take place at baseline and after 4, 8, and 12 months. Assessments will include completing diagnostic interviews and questionnaires, measuring medication adherence through an electronic pill cap, and determining CD4 cell count and viral load (indicators of HIV treatment effectiveness).

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Current diagnosis of depression or prescribed an antidepressant medication with at least some residual symptoms (e.g., clinical global impressions [CGI] scale score of 2 or greater)
* Prescribed a stable regimen of highly active antiretroviral therapy (HAART) for HIV for at least 2 months

Exclusion Criteria:

* Active, untreated, and unstable major mental illness (i.e., untreated psychosis or mania) that would interfere with cognitive behavioral therapy (CBT) treatment for depression
* Diagnosis with any primary psychotic disorder, even if treated
* Treatment with CBT within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
changes in HIV medication adherence, as measured by electronic medication event monitoring system (MEMS) pill-cap scores | Measured at each visit - baseline, interim visits, and after 4, 8, and 12 months
  HIV medication adherence is assessed more frequently during the acute study period (baseline to post-treatment), and then at the follow up major visits.

SECONDARY OUTCOMES:
changes in Severity of depression, as assessed on the Montgomery-Asberg Depression Rating Scale (MADRS) by a blinded independent assessor | Measured at baseline and after 4, 8, and 12 months
changes in depression, as measured by the blinded assessor CGI rating | Measured at baseline and after 4, 8, and 12 months
changes in RNA viral load | Measured at baseline and after 4, 8, and 12 months
changes in CD4 cell count | Measured at baseline and after 4, 8, and 12 months
changes in self-reported depression (CESD) | Measured at each visit
  This is measured more frequently during the acute phase (pretreatment to post-treatment) then at the follow up assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Safren, PhD, Principal Investigator — Partners HealthCare; C. Andres Bedoya, PhD, Study Director — Partners HealthCare
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Fenway Community Health Center, Boston, Massachusetts
  - Butler Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island